CLINICAL TRIAL: NCT04207151
Title: Expanding PrEP By Embedding Unannounced SNAPS Navigators in High Sexually Transmitted Infection (STI) Testing Clinical Sites
Brief Title: Expanding PrEP By Embedding Unannounced SNAPS Navigators in High STI Testing Clinical Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-00060
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hiv; Sexually Transmitted Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants will receive HIV and STI testing, clinical monitoring, client centered counseling and PrEP prescriptions as standard of care, this includes scheduled visits every three months.
- Pre- and Post- SNAPS intervention (Experimental): In addition to the standard of care treatment, approximately twenty subjects will be selected for interview pre- and post-SNAPS intervention to assess PrEP facilitators and barriers for uptake. Participants of interest include cis- and trans-women, for which there is limited data regarding PrEP and HIV prevention.
  Interventions: Behavioral: SNAPS intervention

INTERVENTIONS:
Behavioral: SNAPS intervention — The intervention is multi-level yet, targets the "weakest chains in the link" of PrEP initiation at safety-net hospitals designed for scalability, sustainability, and implementability across a wide range of settings. It consists of Surveillance by STI testing, Navigation by unannounced patient navigators to the Sexual Health Clinic (SHC), Accelerated follow-up with providers with PrEP expertise, Point-of-care PrEP counseling and laboratory testing, and Seamless, consistent, longitudinal, comprehensive care (SNAPS). SNAPS will selectively target those care settings where PrEP prescribing is particularly rare or absent (eg, OB/GYN). Study team will utilize a quasi- experimental design to compare rates of PrEP uptake overall, PrEP initiation in disproportionately-impacted groups, and PrEP retention pre-versus post-initiation of SNAPS, controlling for secular trends.
  Arms: Pre- and Post- SNAPS intervention

SUMMARY:
The goal of this study is to assess the impact of an intervention, known as SNAPS, to expand Preexposure Prophylaxis (PrEP) prescriptions at Health + Hospitals (H+H)/Bellevue. In addition, evaluating whether this intervention, ie SNAPS, helps patients get on PrEP and stay on PrEP to prevent STIs like HIV. PrEP is a medication that needs to be taken on a regular basis in order to be effective to prevent HIV transmission.

DETAILED DESCRIPTION:
The objective of the investigator's proposal is to evaluate the effectiveness of an intervention to (1) increase PrEP initiation overall, (2) increase uptake among groups disproportionately impacted by the HIV pandemic, and (3) to preserve high PrEP retention while expanding use. In addition, the proposal includes innovative secondary outcomes of (4) identifying barriers and facilitators of PrEP use that may be unique to urban safety-net populations, and (5) estimating the HIV infections averted due to greater PrEP uptake from the intervention.

The intervention is multi-level yet, targets the "weakest chains in the link" of PrEP initiation at safety-net hospitals designed for scalability, sustainability, and implementability across a wide range of settings. It consists of Surveillance by STI testing, Navigation by unannounced patient navigators to the Sexual Health Clinic (SHC), Accelerated follow-up with providers with PrEP expertise, Point-of-care PrEP counseling and laboratory testing, and Seamless, consistent, longitudinal, comprehensive care (SNAPS).

ELIGIBILITY:
Inclusion Criteria:

Historical comparison group:

* all adults ≥18 years of age prescribed PrEP at H+H/Bellevue one year prior to SNAPS intervention initiation.

Prospective group:

* all patients will be considered for study participation who are accessing care at H+H/Bellevue ≥ 18 years of age,
* have unknown HIV status,
* requesting STI testing/treatment or inquiring about PrEP or PEP in the ED or urgent care, OB/GYN, and Dermatology clinics.

Exclusion Criteria:

* patients who are HIV positive
* refuse consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Change in PrEP prescriptions | Visits 3 months, 6 months, and 12 months
  Change in rate of PrEP prescriptions at H+H/Bellevue among those in care for 1-year before study period and during 1-year study period by gender, race/ethnicity, age, insurance type, and preferred language.
Change in the knowledge of HIV | Visit baseline, Visit 12 months
  Through pre and post qualitative interviews, the perceived HIV risk, knowledge and attitudes regarding PrEP, and facilitators and barriers regarding PrEP use will be analyzed.
Change in the number of HIV cases | Visit 12 months
  The number of HIV cases averted and distribution of these cases among disproportionately-impacted groups will be assessed to determine if intervention is effective

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pitts, MD, Principal Investigator — New York University
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only by NYU/Bellevue researchers